CLINICAL TRIAL: NCT05934136
Title: My Healthy Brain: A Group-Based Lifestyle Intervention to Modify Early Risk of Dementia in Older Adults
Brief Title: Brain Health Program for Older Adults With Subjective Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ryan A., Mace, PHD, Staff Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P001770
Record Dates: First submitted 2023-06-22; First posted 2023-07-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Memory Loss (Excluding Dementia); Healthy Lifestyle; Risk Reduction Behavior
MeSH Terms: conditions — Memory Disorders; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Healthy Brain 1 (Experimental): My Healthy Brain 1 is an 8-week group program delivered via 90-minute Zoom meetings led by a clinical psychologist. It provides education on the link between dementia and lifestyle factors, including poor exercise, sleep, diet/nutrition, mental and social stimulation, alcohol, and smoking. My Healthy Brain 1 participants learn evidence-based mindfulness and behavior change skills to address common barriers to healthy habits, such as stress and setting achievable goals. My Healthy Brain 1 participants wear an activity watch to monitor lifestyle changes during the program.
  Interventions: Behavioral: My Healthy Brain 1
- My Healthy Brain 2 (Active Comparator): My Healthy Brain 2 condition controls for the effect of time spent and support/feedback from the group and interventionist. Participants in My Healthy Brain 2 will receive education on lifestyle, brain health, and cognitive decline symptoms in addition to usual care as determined by their medical team. Each weekly session will focus on a different topic: 1) lifestyle and brain health, 2) physical activity, 3) sleep, 4) nutrition, 5) medical adherence, 6) cognitive health, 7) social support, and 8) a program overview. My Healthy Brain 2 is conducted in the same format as My Healthy Brain 1 (8 weekly Zoom sessions, 90 minutes each), but does not include behavior change strategies. My Healthy Brain 2 participants wear an activity watch to monitor lifestyle changes during the program.
  Interventions: Behavioral: My Healthy Brain 2

INTERVENTIONS:
Behavioral: My Healthy Brain 1 — My Healthy Brain 1 is an 8-week group program delivered via 90-minute Zoom meetings led by a clinical psychologist. It provides education on the link between dementia and lifestyle factors, including poor exercise, sleep, diet/nutrition, mental and social stimulation, alcohol, and smoking. My Healthy Brain 1 participants learn evidence-based mindfulness and behavior change skills to address common barriers to healthy habits, such as stress and setting achievable goals. My Healthy Brain 1 participants wear an activity watch to monitor lifestyle changes during the program.
  Arms: My Healthy Brain 1
Behavioral: My Healthy Brain 2 — My Healthy Brain 2 condition controls for the effect of time spent and support/feedback from the group and interventionist. Participants in My Healthy Brain 2 will receive education on lifestyle, brain health, and cognitive decline symptoms in addition to usual care as determined by their medical team. Each weekly session will focus on a different topic: 1) lifestyle and brain health, 2) physical activity, 3) sleep, 4) nutrition, 5) medical adherence, 6) cognitive health, 7) social support, and 8) a program overview. My Healthy Brain 2 is conducted in the same format as My Healthy Brain 1 (8 weekly Zoom sessions, 90 minutes each), but does not include behavior change strategies. My Healthy Brain 2 participants wear an activity watch to monitor lifestyle changes during the program.
  Arms: My Healthy Brain 2

SUMMARY:
The investigators will compare two brain health programs in older adults with subjective cognitive decline and lifestyle risk factors for dementia. The primary aim of the study is to determine the credibility, expectancy, feasibility, acceptability, appropriateness, fidelity, and satisfaction of the programs.

DETAILED DESCRIPTION:
The investigators aim to promote brain health by reducing lifestyle risk factors for dementia in older adults with subjective cognitive decline (SCD). This study is a pilot randomized control trial (RCT) comparing two virtual lifestyle programs, My Healthy Brain 1 and My Healthy Brain 2. Eligible older adults include: age ≥ 60, self-reported worry about changes in memory or thinking, and risk factors for dementia (determined by the Cardiovascular Risk Factors, Aging, and Incidence of Dementia score ≥ 6). Participants will be randomized to one of two groups (My Healthy Brain 1 or My Healthy Brain 2) and will complete 8 weekly 90-minute sessions via Zoom delivered by a clinical psychologist. Each session will focus on a different topic relevant to brain health (e.g. physical activity, sleep, etc.). The primary aim of the study is to determine the credibility, expectancy, feasibility, acceptability, appropriateness, fidelity, and satisfaction of the programs. The investigators will also explore improvements in cognition, lifestyle behaviors (physical activity, sleep, nutrition, alcohol and tobacco use, social functioning), depression, anxiety, and mindfulness assessed at baseline, post-intervention, and 6 month follow-up. All participants will wear a watch to monitor changes in lifestyle during the program.

ELIGIBILITY:
Inclusion Criteria:

* Concerns about memory or thinking (subjective cognitive decline, SCD) aged 60 or older
* Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) ≥ 6
* Telephone Interview for Cognitive Status-41 ≥ 31
* Functional Assessment Questionnaire < 9
* English fluency/literacy
* Ability and willingness to participate via live video
* No self-reported safety issues with initiating lifestyle changes during the study

Exclusion Criteria:

* Mild cognitive impairment, dementia, or neurodegenerative disease
* Psychotropic medications (e.g., antidepressant) change in the last 3 months
* Psychosis, uncontrolled bipolar disorder or substance dependence; schizophrenia or schizoaffective disorder
* Current self-report of suicidal ideation
* Serious medical illness expected to worsen in 6 months (e.g., cancer)
* Use of digital monitoring device (e.g., Fitbit) in the last 3 moths AND unwillingness to stop using personal digital monitoring device for duration of program
* Mindfulness or mind-body practice (> 45 min/wk) focused on lifestyle, cognitive-behavioral therapy in < 3 months, or participation in a lifestyle prevention program (ex: diabetes prevention) in < 3 months
* Average daily step count > 5,000 steps
* More than 30 minutes of exercise daily

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Credibility and Expectancy Questionnaire | 0 Weeks
  Assesses how believable, convincing, and logical patients perceive the treatment to be. Higher scores (min = 3, max = 27) scores indicate greater credibility and expectancy.
Client Satisfaction Questionnaire | 8 Weeks
  Assesses patient satisfaction with the program. Higher total scores (min = 3, max = 12) indicate greater satisfaction.
Rates of Recruitment and Enrollment | 0 Weeks
  We will assess the feasibility of recruiting and enrolling participants into the study by calculating the proportion who agree to participate divided by the total number contacted (≥70% good, ≥ 80% excellent).
Rates of Missing Outcomes Data | 8 Weeks
  We will assess the feasibility of data collection by calculating the proportion of secondary outcomes (cognition and lifestyle) with no missing data divided by the total number collected (≥70% good, ≥ 80% excellent).
Rates of Valid Activity Watch Data (10 or more hours of wear time) | 8 Weeks
  We will assess the feasibility of collecting valid activity watch data by calculating the proportion of participants who wore the watch at least 5 out of 7 days per week for at least 10 or more hours per day, divided by the total number of days in the program (≥ 70% good, ≥ 80% excellent).
Rates of Ecological Momentary Assessment (EMA) Data | 8 Weeks
  We will assess the feasibility of collecting ecological momentary assessment (EMA) of daily mindfulness practice by calculating the proportion of participants who complete at least 5 out of 7 daily surveys per week (≥ 70% good, ≥ 80% excellent).
Rates of Treatment Completion | 8 Weeks
  We will assess the acceptability of treatment by calculating the proportion of participants who attend ≥ 6/8 treatment sessions (≥ 70% good, ≥ 80% excellent).
Rates of Therapist Fidelity to Intervention Procedures | 8 Weeks
  We will assess the fidelity of therapists to the intervention procedures by calculating the proportion of sessions with completed audio recordings, progress notes, and checklist with 100% of content delivered divided by the total number of sessions (≥ 75% good, 100% excellent).
Rates of Staff Fidelity to Study Procedures | 8 Weeks
  We will assess the fidelity of staff to the study procedures by counting the frequency of protocol deviations (<5 deviations good, 0 deviations excellent).
Modified Patient Global Impression of Change at 8 weeks | 8 Weeks
  The proportion of participants who report perceived improvements in cognitive function, lifestyle, and emotional well-being outcomes (1=Very Much Worse, 7=Very Much Improved).
Rate of Adverse Events | 8 Weeks
  We will assess the safety of the study by founding the number and severity of adverse events (mild in ≤ 10% of participants = good, none = excellent).

SECONDARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 0 Weeks, 8 Weeks, 6 Months
  A comprehensive test of five cognitive domains (immediate memory, visuospatial/constructional, language, attention, and delayed memory) and global cognition. Higher Z and Index Scores indicate greater cognitive functioning on each domain.
Cognitive Function Instrument | 0 Weeks, 8 Weeks, 6 Months
  14-item self-report of cognitive and functional status. Higher total scores (min=0, max=14) indicate greater subjective cognitive complaints.
Change in Step Count | 0 Weeks, 8 Weeks, 6 Months
  Activity watch change in steps count during the 7 days preceding baseline assessment, throughout the intervention period, and 7 days at 6-month follow-up. Higher step count totals indicate greater physical activity (walking).
PROMIS Physical Function | 0 Weeks, 8 Weeks, 6 Months
  8-item self-report of daily functioning. Higher T scores (mean = 50, sd = 10) indicate greater physical function.
Change in Total Sleep Time | 0 Weeks, 8 Weeks, 6 Months
  Activity watch change in total sleep time during the 7 days preceding baseline assessment, throughout the intervention period, and 7 days at 6-month follow-up. Higher total minutes indicate greater sleep time.
Pittsburgh Sleep Quality Index | 0 Weeks, 8 Weeks, 6 Months
  9-item self-report of sleep patterns and overall quality. Higher total scores (min=0, max=21) indicate greater sleep disturbance (>5 = clinically significant).
Mediterranean Eating Pattern for Americans Screener | 0 Weeks, 8 Weeks, 6 Months
  16-item self-report of adherence to Mediterranean dietary recommendations. Higher total scores (min=0, max=21) indicate greater intake/adherence of Mediterranean foods.
PROMIS Alcohol Use | 0 Weeks, 8 Weeks, 6 Months
  7-item self-report of at-risk drinking. Higher T scores (mean = 50, sd = 10) indicate greater problematic alcohol use.
CDC Other Tobacco Product Use Questions | 0 Weeks, 8 Weeks, 6 Months
  2-item self-report of the frequency and use of 6 common tobacco products (1=Less than once a month, 5=Daily or almost daily).
PROMIS Satisfaction with Social Roles and Activities | 0 Weeks, 8 Weeks, 6 Months
  8-item self-report measure of satisfaction of performing usual social roles and activities. Higher T scores (mean = 50, sd = 10) indicate greater satisfaction with social roles and activities.

OTHER OUTCOMES:
Measure of Cognitive Activities | 0 Weeks, 8 Weeks, 6 Months
  10-item self-report measure of frequency of certain cognitive activities (e.g. reading newspapers, playing music, etc). Higher total scores (min=0, max=10) indicate greater participation in cognitively stimulating activities.
Memory Compensation Questionnaire | 0 Weeks, 8 Weeks, 6 Months
  13-item self-report that assesses the variety and extent to which an individual compensates for actual or perceived memory losses. Higher total scores (min=0, max=65) indicate greater utilization of memory compensation strategies.
Godin Leisure-Time Exercise Questionnaire | 0 Weeks, 8 Weeks, 6 Months
  3-item self-report of weekly engagement in light, moderate, and vigorous physical activities. Higher average scores indicate greater engagement in total physical activity.
Social Engagement and Activities Questionnaire | 0 Weeks, 8 Weeks, 6 Months
  10-item self-report measure of perceived frequency of specific social activities. Higher total scores (min=0, max=50) indicate greater participation in socially engaging activities.
PROMIS Loneliness | 0 Weeks, 8 Weeks, 6 Months
  5-item self-report of perceived loneliness. Higher T scores (mean = 50, sd = 10) indicate greater perceived loneliness.
PROMIS Depression and Anxiety | 0 Weeks, 8 Weeks, 6 Months
  4-item self-reports of each construct. Higher T scores (mean = 50, sd = 10) indicate greater depression and anxiety.
Applied Mindfulness Process Scale | 0 Weeks, 8 Weeks, 6 Months
  15-item self-report of using basic mindfulness principles. Higher total scores (min=0, max=60) indicate greater utilization in daily mindfulness activities.
Cognitive Control and Flexibility Questionnaire | 0 Weeks, 8 Weeks, 6 Months
  13-item self-report of control over unwanted experiences. Higher total scores (min=13, max=52) indicate greater daily utilization of cognitive control and flexibility.
Emotion Regulation Questionnaire | 0 Weeks, 8 Weeks, 6 Months
  10-item self-report of emotion regulation strategies. Higher total scores (min=10, max=70) indicate greater utilization of emotional regulation strategies.
Motivation to Change Lifestyle and Health Behaviours for Dementia Risk Reduction | 0 Weeks, 8 Weeks, 6 Months
  27-item self report of motivation and perceived self-efficacy of lifestyle and health behavior change for dementia risk reduction. Higher total scores (min=27, max=135) indicate greater motivation to alter lifestyle factors and health behaviors to reduce risk of dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mace RA, Hopkins SW, Reynolds GO, Vranceanu AM. My Healthy Brain: Rationale and Case Report of a Virtual Group Lifestyle Program Targeting Modifiable Risk Factors for Dementia. J Clin Psychol Med Settings. 2022 Dec;29(4):818-830. doi: 10.1007/s10880-022-09843-2. Epub 2022 Jan 25. PMID 35079948
- [Result] Mace RA, Greenberg J, Stauder M, Reynolds G, Vranceanu AM. My Healthy Brain: a multimodal lifestyle program to promote brain health. Aging Ment Health. 2022 May;26(5):980-991. doi: 10.1080/13607863.2021.1904828. Epub 2021 Mar 30. PMID 33784902
- [Result] Mace RA, Popok PJ, Hopkins SW, Fishbein NS, Vranceanu AM. Adaptation and virtual feasibility pilot of a mindfulness-based lifestyle program targeting modifiable dementia risk factors in older adults. Aging Ment Health. 2023 Apr;27(4):695-707. doi: 10.1080/13607863.2022.2032600. Epub 2022 Feb 1. PMID 35100922
- [Derived] Mace RA, Law ME, Cohen JE, Ritchie CS, Okereke OI, Hoeppner BB, Brewer JA, Bartels SJ, Vranceanu AM; My Healthy Brain Team. A Mindfulness-Based Lifestyle Intervention for Dementia Risk Reduction: Protocol for the My Healthy Brain Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2024 Nov 21;13:e64149. doi: 10.2196/64149. PMID 39571150